CLINICAL TRIAL: NCT04137952
Title: The Use of Neuro-cognitive Strategies to Power Generalization Effect After Short-term Postural Training for Older Adults
Brief Title: Short-term Postural Training for Older Adults
Acronym: P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MOST 108-2314-B-006-071 -
Record Dates: First submitted 2019-10-20; First posted 2019-10-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging; Balance
Keywords: Posture training, Motor generalization, Aging, Cognition, High-density electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- deterministic visual error gain (Experimental): Day1(Pretest):
  1. stabilometer stance, 3 times/1 min
  2. air pillow stance, 3 time/30 sec
  3. poture-supraposture dual task, 3 times/1 min
  Day2 to Day5:
  1. Exp.group:27 times of posture tracking with high visual error gain.
  2. Control group:27 times of posture training with normal visual error gain.
  Day6 (Posttest):
  1. stabilometer stance, 3 times/1 min
  2. air pillow stance, 3 time/30 sec
  3. poture-supraposture dual task, 3 times/1 min
  Interventions: Behavioral: size of error visual feedback
- stochastic visual noise (Experimental): Day1(Pretest):
  1. stabilometer stance, 3 times/1 min
  2. air pillow stance, 3 time/30 sec
  3. poture-supraposture dual task, 3 times/1 min
  Day2 to Day5:
  1. Exp.group A:27 times of posture training with posture tracking signal-to-noise ratio=2:1.
  2. Exp.group B:27 times of posture training with posture tracking signal-to-noise ratio=4:1.
  3. Control group:27 times of posture training with normal visual error gain.
  Day6(Posttest):
  1. stabilometer stance, 3 times/1 min
  2. air pillow stance, 3 time/30 sec
  3. poture-supraposture dual task, 3 times/1 min
  Interventions: Behavioral: size of error visual feedback
- intermittent visual gain (Experimental): Day1 (Pretest):
  1. stabilometer stance with wearing flash glasses (low frequency with opaque ratio 50%), 4 times/45 sec
  2. stabilometer stance with wearing flash glasses (high frequency with opaque ratio 50%), 4 times/45 sec.
  3. stabilometer stance with wearing flash glasses (clear), 4 times/45 sec
  4. air pillow stance, 8 times/1 min
  Day2 (training section):
  1. Exp. group:Posture tracking with wearing flash glasses (low frequency with opaque ratio 50%), 12 times/45 sec.
  2. Control group:Posture tracking with wearing flash glasses (clear), 12 times/45 sec.
  Day3 (Posttest):
  1. stabilometer stance with wearing flash glasses (low frequency with opaque ratio 50%), 4 times/45 sec
  2. stabilometer stance with wearing flash glasses (high frequency with opaque ratio 50%), 4 times/45 sec
  3. stabilometer stance with wearing flash glasses (clear), 4 times/45 sec
  4. air pillow stance, 8 times/1 min
  Interventions: Behavioral: size of error visual feedback

INTERVENTIONS:
Behavioral: size of error visual feedback — The strategies are expected to enhance opportunities of error experience and motor exploration via modified visual feedback, underlying facilitations of attentional resource and error-related neural networks.
  Other Names: virtual uncertainness of motor goals; stroboscopic vision

SUMMARY:
Generalization refers to skill transfer under various working spaces following motor practice. The extent of generalization effect links causal to in-depth recognition of error properties during motor practice. Idiom says "imperfect practice makes perfect". It could be beneficial for the elderly to gain superior capacity of balance transfer skill under the short-term productive failure learning environments. In contrast to traditional visual feedback that uses error avoidance training to optimize target balance task, the present 3-year proposal is to propose three potential neuro-cognitive strategies to improve motor skill transfer following stabilometer training. The strategies are expected to enhance opportunities of error experience and motor exploration via modified visual feedback, underlying facilitations of attentional resource and error-related neural networks. In the first year, the neuro-cognitive strategy for balance practice is progressive augmentation of visual error size to improve balance skill transfer. In the second year, the neuro-cognitive strategy for balance practice is visual feedback with virtual uncertainness of motor goal. In the third year, the neuro-cognitive strategy for balance practice is stroboscopic vision. EEG and central of pressure will be processed with non-linear approaches. Graph theory will characterize EEG functional connectivity and brain network efficiency regarding to brain mechanisms for practice-related leaning transfer. Trajectories of central of pressure will be analyzed with stabilogram diffusion analysis to reveal behavior mechanisms for practice-related variations in feedback and feedforward process for error corrections.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years old healthy older adults without a history of falls.
* Able to understand and give informed consent.
* The Mini-Mental State Examination test score above 25-30.
* Lower limb muscle strength is evaluated as G grade
* The corrected visual acuity was within the normal range.

Exclusion Criteria:

* Any known history of mental illness
* Any neuromuscular or degenerative neurological disease(ex:stroke、SCI、TBI...etc)
* Any known history of cerebral cerebellar disease or intracranial metal implants.
* Weak of hearing or wearing a hearing aid

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
EEG graph analysis | through study completion, an average of 1 year
  Graph theory will characterize EEG functional connectivity and brain network efficiency regarding to brain mechanisms for practice-related leaning transfer.

SECONDARY OUTCOMES:
stabilogram diffusion analysis of central of pressure | through study completion, an average of 1 year
  Trajectories of central of pressure will be analyzed with stabilogram diffusion analysis to reveal behavior mechanisms for practice-related variations in feedback and feedforward process for error corrections.
root mean sqaure error of stabilometer | through study completion, an average of 1 year
  The root-mean-square value of the tracking trajectory of stabilometer and the target signal.

CONTACTS AND LOCATIONS:
Overall Officials: Hwang Ing-Shiou, Phd, Study Chair — NCKU, Institute of Allied Health Sciences
Locations (1):
- National Chen Kong University Hospital, Taian, Eastern District, Taiwan

IPD SHARING:
Plan to Share IPD: No